CLINICAL TRIAL: NCT03364946
Title: High Flow Nasal Cannula Technique in Iberoamerica
Brief Title: High Flow Therapy in ICUs Across Ibero America
Acronym: T-Calfi
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Leopoldo Ferrer, Principal investigator, Fundación Santa Fe de Bogota
Other Study IDs: CCEI-7327-2017
Record Dates: First submitted 2017-11-20; First posted 2017-12-07 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Nasal High Flow Therapy; Intensive Care Unit; Ventilatory Failure; Hypoxia; Hypercapnic Respiratory Failure
MeSH Terms: conditions — Hypoventilation; Hypoxia; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High Nasal Flow Therapy: Every patient in the ICU that requires High Nasal Flow Therapy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention, observational study

SUMMARY:
The study aims to describe the use of Nasal High Flow (NHF) in the intensive care units of participating centers in Iberoamerica. It will describe the indications for the use, the clinical outcome of patients , and the therapeutic failure of NHF therapy in patients staying in an intensive care unit in the participant centers in Iberoamerica.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Admitted to medical or surgical ICU
* Requirement of high nasal flow therapy

Exclusion Criteria:

* Post-extubation failure
* Patient unable to protect airway
* Diagnosed shock
* Glasgow equal or under 8

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old, admitted to an ICU in the reference centers in Iberoamerica, requiring the use of high nasal flow therapy
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Hypoxemia | 15 days
  PO2 under 60mmHg, or SatO2 under 80%; that leads to the instauration of invasive ventilation
Tachypnea | 15 days
  Respiratory rate over 20; that leads to the instauration of invasive ventilation
Hypercapnia | 15 days
  PCO2 over 55mmHg; that leads to the instauration of invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo E Ferrer, MD, Principal Investigator — Fundación Santa Fe de Bogotá
Locations (9):
- Colombia (4):
  - Fundación Santa Fe de Bogotá, Bogotá, Bogota D.C.
  - Hospital Departamental de Nariño, Nariño, Pasto
  - Medicina Intensiva del Tolima, Ibagué, Tolima Department
  - Clinica Reina Sofia, Bogotá
- Instituto Nacional del Cáncer Rosa Emilia Sánchez Pérez de Tavarez (INCART), Santo Domingo, Dominican Republic
- Fundación Medica Sur, Mexico City, Mexico City, Mexico
- Spain (3):
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - MD Anderson Cancer Center, Madrid
  - Hospital Ramon y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to external researchers prior to publication